CLINICAL TRIAL: NCT01361009
Title: Safety of Pramipexole Monotherapy or Combination Therapy in Chinese Patients With Parkinson¿s Disease: a 12 Week Post Marketing Surveillance
Brief Title: a PMS on Safety Profile of Pramipexole in Chinese Parkinson Disease Patients
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.682
Record Dates: First submitted 2011-05-23; First posted 2011-05-26 (Estimated); Results first posted 2013-08-30 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2013-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- pramipexole group: It's a open-label, non-intervention,observation post marketing surveillance to observe the safety and efficacy of pramipexole in real world.
  Interventions: Drug: pramipexole

INTERVENTIONS:
Drug: pramipexole — as prescibed by the investigator

SUMMARY:
This is an open-label, multicenter, non-interventional, prospective observational study. we collect the safety information of pramipexole over 12w treatment. Parkinson disease patients with different severity who have already used pramipexole could be observed in this study. In the whole observation period, treatment decision was determined by physician and patient completely. The safety endpoint is AE(Adverse Event), SAE(Serious Adverse Event), patient withdraw, laboratory test.

DETAILED DESCRIPTION:
Purpose:

ELIGIBILITY:
Inclusion criteria:

1. Diagnosed as idiopathic PD (Parkinson' disease) according to UK brain bank criteria
2. Age: from 30 to 75 years old
3. Stage I-IV of revised Hoehn-Yahr standards
4. With current use of pramipexole
5. Informed consent signed by every subject

Exclusion criteria:

1. Diagnosis of Parkinson¿s syndrome
2. Current use of psychotolytic medications
3. Allergic to pramipexole or any other ingredient of pramipexole
4. Female patients in pregnancy and lactation
5. Patients who were participating in other clinical studies by signing relevant informed consent or who received other investigational drugs within 30 days prior to the study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3000
Sampling Method: Probability Sample
Enrollment: 2017 (Actual)
Dates: Start 2011-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (103):
- China (103):
  - Boehringer Ingelheim Investigational Site 54, Beijing
  - Boehringer Ingelheim Investigational Site 55, Beijing
  - Boehringer Ingelheim Investigational Site 56, Beijing
  - Boehringer Ingelheim Investigational Site 57, Beijing
  - Boehringer Ingelheim Investigational Site 58, Beijing
  - Boehringer Ingelheim Investigational Site 59, Beijing
  - Boehringer Ingelheim Investigational Site 60, Beijing
  - Boehringer Ingelheim Investigational Site 61, Beijing
  - Boehringer Ingelheim Investigational Site 62, Beijing
  - Boehringer Ingelheim Investigational Site 63, Beijing
  - Boehringer Ingelheim Investigational Site 64, Beijing
  - Boehringer Ingelheim Investigational Site 65, Beijing
  - Boehringer Ingelheim Investigational Site 66, Changchun
  - Boehringer Ingelheim Investigational Site 67, Changchun
  - Boehringer Ingelheim Investigational Site 12, Changsh
  - Boehringer Ingelheim Investigational Site 13, Changsh
  - Boehringer Ingelheim Investigational Site 14, Changsh
  - Boehringer Ingelheim Investigational Site 15, Changsh
  - Boehringer Ingelheim Investigational Site 16, Changsh
  - Boehringer Ingelheim Investigational Site 94, Chendu
  - Boehringer Ingelheim Investigational Site 95, Chendu
  - Boehringer Ingelheim Investigational Site 100, Chongqing
  - Boehringer Ingelheim Investigational Site 101, Chongqing
  - Boehringer Ingelheim Investigational Site 97, Chongqing
  - Boehringer Ingelheim Investigational Site 98, Chongqing
  - Boehringer Ingelheim Investigational Site 99, Chongqing
  - Boehringer Ingelheim Investigational Site 71, Dalian
  - Boehringer Ingelheim Investigational Site 72, Dalian
  - Boehringer Ingelheim Investigational Site 79, Daqing
  - Boehringer Ingelheim Investigational Site 35, Fuzhou
  - Boehringer Ingelheim Investigational Site 36, Fuzhou
  - Boehringer Ingelheim Investigational Site 37, Fuzhou
  - Boehringer Ingelheim Investigational Site 80, Guangzhou
  - Boehringer Ingelheim Investigational Site 81, Guangzhou
  - Boehringer Ingelheim Investigational Site 82, Guangzhou
  - Boehringer Ingelheim Investigational Site 83, Guangzhou
  - Boehringer Ingelheim Investigational Site 84, Guangzhou
  - Boehringer Ingelheim Investigational Site 85, Guangzhou
  - Boehringer Ingelheim Investigational Site 86, Guangzhou
  - Boehringer Ingelheim Investigational Site 87, Guangzhou
  - Boehringer Ingelheim Investigational Site 88, Guangzhou
  - Boehringer Ingelheim Investigational Site 89, Guangzhou
  - Boehringer Ingelheim Investigational Site 90, Guangzhou
  - Boehringer Ingelheim Investigational Site 91, Guangzhou
  - Boehringer Ingelheim Investigational Site 77, Haerbin
  - Boehringer Ingelheim Investigational Site 78, Haerbin
  - Boehringer Ingelheim Investigational Site 28, Hangzhou
  - Boehringer Ingelheim Investigational Site 29, Hangzhou
  - Boehringer Ingelheim Investigational Site 30, Hangzhou
  - Boehringer Ingelheim Investigational Site 31, Hangzhou
  - Boehringer Ingelheim Investigational Site 32, Hangzhou
  - Boehringer Ingelheim Investigational Site 38, Hefei
  - Boehringer Ingelheim Investigational Site 39, Jinan
  - Boehringer Ingelheim Investigational Site 40, Jinan
  - Boehringer Ingelheim Investigational Site 96, Luzhou
  - Boehringer Ingelheim Investigational Site 53, Nanchang
  - Boehringer Ingelheim Investigational Site 44, Nanjing
  - Boehringer Ingelheim Investigational Site 45, Nanjing
  - Boehringer Ingelheim Investigational Site 46, Nanjing
  - Boehringer Ingelheim Investigational Site 47, Nanjing
  - Boehringer Ingelheim Investigational Site 48, Nanjing
  - Boehringer Ingelheim Investigational Site 49, Nantong
  - Boehringer Ingelheim Investigational Site 43, Qingdao
  - Boehringer Ingelheim Investigational Site 17, Shanghai
  - Boehringer Ingelheim Investigational Site 18, Shanghai
  - Boehringer Ingelheim Investigational Site 19, Shanghai
  - Boehringer Ingelheim Investigational Site 20, Shanghai
  - Boehringer Ingelheim Investigational Site 21, Shanghai
  - Boehringer Ingelheim Investigational Site 22, Shanghai
  - Boehringer Ingelheim Investigational Site 23, Shanghai
  - Boehringer Ingelheim Investigational Site 24, Shanghai
  - Boehringer Ingelheim Investigational Site 25, Shanghai
  - Boehringer Ingelheim Investigational Site 26, Shanghai
  - Boehringer Ingelheim Investigational Site 27, Shanghai
  - Boehringer Ingelheim Investigational Site 92, Shantou
  - Boehringer Ingelheim Investigational Site 73, Shenyang
  - Boehringer Ingelheim Investigational Site 74, Shenyang
  - Boehringer Ingelheim Investigational Site 75, Shenyang
  - Boehringer Ingelheim Investigational Site 76, Shenyang
  - Boehringer Ingelheim Investigational Site 93, Shenzhen
  - Boehringer Ingelheim Investigational Site 2, Shijiazhuang
  - Boehringer Ingelheim Investigational Site 3, Shijiazhuang
  - Boehringer Ingelheim Investigational Site 6, Shiyan
  - Boehringer Ingelheim Investigational Site 51, Suzhou
  - Boehringer Ingelheim Investigational Site 52, Suzhou
  - Boehringer Ingelheim Investigational Site 1, Taiyuan
  - Boehringer Ingelheim Investigational Site 68, Tianjin
  - Boehringer Ingelheim Investigational Site 69, Tianjin
  - Boehringer Ingelheim Investigational Site 70, Tianjin
  - Boehringer Ingelheim Investigational Site 41, Weifang
  - Boehringer Ingelheim Investigational Site 33, Wenzhou
  - Boehringer Ingelheim Investigational Site 10, Wuhan
  - Boehringer Ingelheim Investigational Site 11, Wuhan
  - Boehringer Ingelheim Investigational Site 7, Wuhan
  - Boehringer Ingelheim Investigational Site 8, Wuhan
  - Boehringer Ingelheim Investigational Site 9, Wuhan
  - Boehringer Ingelheim Investigational Site 50, Wuxi
  - Boehringer Ingelheim Investigational Site 102, Xi'an
  - Boehringer Ingelheim Investigational Site 103, Xi'an
  - Boehringer Ingelheim Investigational Site 34, Xiamen
  - Boehringer Ingelheim Investigational Site 42, Yantai
  - Boehringer Ingelheim Investigational Site 4, Zhengzhou
  - Boehringer Ingelheim Investigational Site 5, Zhengzhou

RESULTS

PARTICIPANT FLOW:
Groups:
- Pramipexole Goup: An open-label, non-controlled, non-interventional, observational post marketing surveillance to observe the safety and efficacy of pramipexole in real world.
Period: Overall Study
Arm/Group | Pramipexole Goup
Started | 2017
Completed | 1901
Not Completed | 116
Not completed — Protocol Violation | 116

BASELINE CHARACTERISTICS:
Arm/Group | Pramipexole Goup
Number analyzed (Participants) | 2017
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.09 (9.67)
Gender [Number; unit: Number of participants] — The data of gender in three patients was missing
  Number of participants
    Female | 840
    Male | 1174
Course of Parkinson's disease [Median (Inter-Quartile Range); unit: years] — Course of Parkinson's disease is the length of time that participants had Parkinson's Disease prior to study enrollment.
  years | 3 (2.5) [2 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of AE/SAE
Description: The percentage of adverse events or serious adverse events occurring under Pramipexole mono- or combination therapy with other medication in this study.
Time Frame: 12 weeks
Population: There were 2017 patients in the safety analysis set (SAS). SAS includes the patients who took drug at least once and had safety data. In this study, 2017 patients were recruited, who have been using pramipexole before the enrollment.
Measure: Number; unit: Percentage of participants
Arm/Group | Pramipexole Goup
Number analyzed (Participants) | 2017
Percentage of participants | 5.16

2. Secondary Outcome: Patient Global Impression(PGI) at Visit 1(Baseline) and Visit 3(at the End of Study)
Description: Patient Global Impression (PGI) scale, ranging from 1 (excellent) to 7 (extremely poor), including 1(excellent), 2(very good), 3(good), 4(no change), 5(poor), 6(very poor) and 7(extremely poor).
Time Frame: Baseline (Visit 1) and 12 weeks (Visit 3)
Population: There were 1891 patients in full analysis set(FAS). FAS includes all patients who fulfilled the inclusion criteria and exclusion criteria, without missing PGI values at visit 1 and visit 3. In the recruited 2017 patients, 116 patients didn't fully meet the inclusion or exclusion criteria and 10 patients missed PGI data at visit 1 or visit 3.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Pramipexole Goup
Number analyzed (Participants) | 1891
unit on a scale
  Visit 1 | 3.53 (1.23)
  Visit 3 | 2.48 (0.69)

3. Secondary Outcome: The Dosage Related Information of Pramipexole at Baseline
Description: At enrollment, the distribution of patients in 3 pramipexole dosage categories.
Time Frame: baseline
Population: There were 2017 patients in SAS set.
Measure: Number; unit: percentage of patients
Arm/Group | Pramipexole Goup
Number analyzed (Participants) | 2017
percentage of patients
  dosage < 0.75mg/d | 84.93
  1.5mg/d > dosage ≥ 0.75mg/d | 12.99
  dosage ≥ 1.5mg/d | 2.08

4. Secondary Outcome: The Dosage Related Information of Pramipexole at the End of Study
Description: At the end of study, the distribution of patients in 3 pramipexole dosage categories.
Time Frame: 12 weeks
Population: There were 2017 patients in SAS set
Measure: Number; unit: percentage of patients
Arm/Group | Pramipexole Goup
Number analyzed (Participants) | 2017
percentage of patients
  dosage < 0.75mg/d | 33.56
  1.5mg/d > dosage ≥ 0.75mg/d | 46.16
  dosage ≥ 1.5mg/d | 20.28

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Pramipexole Goup
Serious Adverse Events (participants affected / at risk) | 0/2017
Other Adverse Events (participants affected / at risk) | 0/2017

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.